CLINICAL TRIAL: NCT02664415
Title: Safety and Therapeutic Efficacy of the Broadly Neutralizing HIV-1 Specific Monoclonal Antibody VRC01 During Analytic Treatment Interruption in Patients Who Initiated Antiretroviral Therapy During Early Acute HIV Infection
Brief Title: Safety and Therapeutic Efficacy of the VRC01 Antibody in Patients Who Initiated Antiretroviral Therapy During Early Acute HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RV 397; 12001 (Registry Identifier: DAIDS-ES Registry Number); NCT03036709 (obsolete NCT alias)
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Human Monoclonal Antibody
MeSH Terms: conditions — HIV Infections | interventions — VRC01 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VRC01 (Experimental): Participants will receive an intravenous (IV) infusion of 40 mg/kg of VRC01 at Week 0 and every 3 weeks until Week 24 or until criteria for resumption of ART are met.
  Interventions: Biological: VRC01
- Placebo for VRC01 (Placebo Comparator): Participants will receive an IV infusion of placebo at Week 0 and every 3 weeks until Week 24 or until criteria for resumption of ART are met.
  Interventions: Biological: Placebo for VRC01

INTERVENTIONS:
Biological: VRC01 — 40 mg/kg; administered IV
  Other Names: VRC-HIVMAB060-00-AB
  Arms: VRC01
Biological: Placebo for VRC01 — Sodium Chloride for Injection 0.9%, USP; administered IV
  Arms: Placebo for VRC01

SUMMARY:
The study will evaluate the safety and therapeutic efficacy of the human monoclonal antibody (mAb) VRC-HIVMAB060-00-AB (VRC01), when administered during analytic treatment interruption (ATI), in adults who began antiretroviral therapy (ART) during early acute HIV infection.

DETAILED DESCRIPTION:
Human monoclonal antibodies (mAbs) may have the potential to treat HIV infection by preventing the spread of the virus. This study will evaluate an experimental mAb known as VRC-HIVMAB060-00-AB (VRC01). The purpose of this study is to evaluate the safety and therapeutic efficacy of VRC01, when administered during analytic treatment interruption (ATI), in adults who began antiretroviral therapy (ART) during early acute HIV infection.

The study will enroll participants from the RV 254 study who were diagnosed during early acute HIV infection and who have been on ART. At study entry, participants will stop taking their antiretroviral (ARV) medications. They will be randomly assigned to receive an intravenous (IV) infusion of VRC01 or placebo at Weeks 0 (study entry), 3, 6, 9, 12, 15, 18, 21, and 24. For 7 days following each infusion, participants will be asked to record and report any symptoms to study researchers.

In addition to the infusion visits, participants will attend follow-up visits for 48 weeks. Study visits may include physical examinations, blood collection, and urine collection. Neurocognitive testing will take place at select study visits. Some participants may take part in optional study procedures including mucosal secretion collection, MRI brain scan, colon biopsy, lymph node biopsy, leukapheresis, and lumbar puncture.

Study staff will monitor participants' HIV throughout the study, and participants will end their participation in the study and restart their ARV medications, if needed.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent or, in the case of illiteracy, witnessed verbal informed consent with documentation of a thumbprint in lieu of a signature.
* Passes Test of Understanding.
* Man or woman aged 20-50 years.
* Initiated on ART during acute HIV infection (Fiebig Stage I to III at RV 254 enrollment).
* Prescribed ART for at least 24 months prior to enrollment.
* HIV-1 RNA less than 50 copies/mL on at least three consecutive measurements within the past 12 months.
* Integrated HIV DNA in peripheral blood mononuclear cells (PBMCs) below the level of detection (1 copy/10^5 PBMCs) within 6 months prior to enrollment.
* Last documented peripheral blood CD4 greater than 400 cells/mm^3 within 3 months prior to enrollment.
* No HIV-related or AIDS-defining illness within 6 months prior to enrollment.
* In general good health.
* Able to participate in study visits.

Female-Specific Criteria:

* Agrees not to become pregnant from the time of study enrollment until the last study visit. If a woman is sexually active and has no history of hysterectomy or tubal ligation or menopause, she must agree to use a prescription birth control method or a barrier birth control method.
* Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on day of enrollment for any women unless she is post-menopause for 24 consecutive months or has undergone a surgical procedure that precludes pregnancy.

Exclusion Criteria:

* Previous receipt of humanized or human monoclonal antibody whether licensed or investigational.
* Ongoing AIDS-related opportunistic infection (including oral thrush).
* Active injection drug use within previous 12 months.
* History of a severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis in the 2 years prior to enrollment.
* History of chronic urticaria requiring daily treatment.
* Physical finding on examination considered indicative of significant disease such as murmur (other than functional), hepatosplenomegaly, or focal neurologic deficit.
* Hypertension that is not well controlled by medication.
* Hepatitis B surface antigen positive at any time in the past.
* Hepatitis C antibody positive at any time in the past.
* Untreated syphilis.
* Estimated glomerular filtration rate (GFR) less than 50 ml/min within the past 90 days.
* Pregnant or breastfeeding.
* Receipt of licensed vaccine or other investigational study agent within 28 days prior to enrollment or past participation in an investigational HIV vaccine study with receipt of active product.
* Current or planned participation in another interventional clinical trial during the study period.
* Chronic or recurrent use of medications that modify host immune response, e.g., oral or parenteral steroids, cancer chemotherapy.
* Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer. Including, but not limited to: diabetes mellitus type I, chronic hepatitis, renal failure; OR clinically significant forms of: drug or alcohol abuse, mental illness, severe asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer.
* Study site employee.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Crowell, MD, PhD, Study Chair — US Military HIV Research Program
Locations (1):
- SEARCH Thai Red Cross AIDS Research Centre Non-Network CRS, Bangkok, Thailand

REFERENCES:
- [Derived] Crowell TA, Colby DJ, Pinyakorn S, Sacdalan C, Pagliuzza A, Intasan J, Benjapornpong K, Tangnaree K, Chomchey N, Kroon E, de Souza MS, Tovanabutra S, Rolland M, Eller MA, Paquin-Proulx D, Bolton DL, Tokarev A, Thomas R, Takata H, Trautmann L, Krebs SJ, Modjarrad K, McDermott AB, Bailer RT, Doria-Rose N, Patel B, Gorelick RJ, Fullmer BA, Schuetz A, Grandin PV, O'Connell RJ, Ledgerwood JE, Graham BS, Tressler R, Mascola JR, Chomont N, Michael NL, Robb ML, Phanuphak N, Ananworanich J; RV397 Study Group. Safety and efficacy of VRC01 broadly neutralising antibodies in adults with acutely treated HIV (RV397): a phase 2, randomised, double-blind, placebo-controlled trial. Lancet HIV. 2019 May;6(5):e297-e306. doi: 10.1016/S2352-3018(19)30053-0. Epub 2019 Apr 15. PMID 31000477

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Thai Red Cross AIDS Research Centre in Bangkok, Thailand. Participants were recruited between 9 August 2016 and 9 January 2017, from ongoing Acute HIV Infection (AHI) cohorts and received ART during AHI via a separately-funded protocol (clinicaltrials.gov NCT00796263).
Pre-assignment Details: Twenty-three participants were enrolled, 4 were withdrawn prior to randomization because of the unavailability of study product in-country, and 19 were randomized with 5 assigned to placebo and 14 to VRC01. One VRC01 recipient experienced severe generalized urticaria during the first study infusion and did not complete the study.
Period: Overall Study
Arm/Group | VRC01 | Placebo for VRC01
Started | 14 | 5
Completed | 13 | 5
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRC01 | Placebo for VRC01 | Total
Number analyzed (Participants) | 13 | 5 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 5 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 32 [21 to 50] | 25 [23 to 48] | 29 [21 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 13 | 5 | 18
HIV-subtype [Count of Participants; unit: Participants]
  CRF01_AE | 8 | 4 | 12
  B | 3 | 1 | 4
  CRF01_AE and B co-infection | 1 | 0 | 1
  CRF01_AE/B/C recombinant | 1 | 0 | 1
Feibig stage at ART initiation [Count of Participants; unit: Participants] — Fiebig stage is a laboratory staging system for primary HIV infection (Fiebig et al).
  Stage I: HIV present in blood samples, only RNA assay positive (RNA+); Stage II: RNA+ and HIV-1 p24 antigen positive (p24+), antibody EIA non-reactive (IgM-); Stage III: RNA+, HIV-1 antigen and HIV IgM-sensitive EIA reactive (IgM+), but Western blot without HIV-a-specific band (WB-) .
  The higher stage refers to the later stage of infection.
  Participants
    I (RNA+, p24-) | 1 | 0 | 1
    II (p24+, IgM-) | 7 | 3 | 10
    III (IgM+, WB-) | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Event
Description: Participants were monitored for up to 10 weeks after the last infusion of VRC01 or placebo
Time Frame: Measured up to 10 weeks after last infusion of VRC01 or placebo
Population: Participants who were randomized to receive VRC01 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 14 | 5
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Sustained Virologic Suppression
Description: Number of participants who sustained virologic control (HIV RNA <50 copies/mL), without indication for ART resumption at week 24.
Time Frame: Measured through 24 weeks after ATI
Population: This is the number of participants who received at least one full dose of VRC01 or placbo, underwent Analytic Treatment Interruption (ATI).
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 13 | 5
Participants | 1 | 0
Statistical Analysis 1: Comparison: VRC01 vs Placebo for VRC01; Test type: Superiority; p = 1.000, Fisher Exact; This is to confirm that the p-value from Fisher's Exact test was 1.000

3. Secondary Outcome: Time to Viral Rebound After Cessation of ART
Description: This is the days from Analytic Treatment Interruption (ATI) to:
  1. HIV RNA >= 20 copies/mL.
  2. HIV RNA >= 1000 copies/mL
Time Frame: Measured from Baseline ATI through ART resumption.
Population: Participants who received at least 1 full dose of VRC01 or Placebo and underwent ATI.
Measure: Median (Full Range); unit: days
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 13 | 5
days
  Time from ATI to HIV-1 RNA >= 20 copies/mL | 29 [9 to 296] | 14 [14 to 29]
  Time from ATI to HIV-1 RNA >= 1000 copies/mL | 33 [13 to 305] | 14 [14 to 32]
Statistical Analysis 1: Comparison: VRC01 vs Placebo for VRC01; A comparison of time from ATI to HIV-1 RNA >= 20 copies/mL between arms; Test type: Superiority; p = 0.051, Log Rank
Statistical Analysis 2: Comparison: VRC01 vs Placebo for VRC01; A comparison of time from ATI to HIV-1 RNA >= 1000 copies/mL between arms; Test type: Superiority; p = 0.01, Log Rank

4. Secondary Outcome: Level of Rebound Viremia After Cessation of ART
Description: This is the HIV-1 RNA levels (copies/mL) at first detection and ART resumption.
Time Frame: Measured from Baseline ATI through ART resumption.
Population: Participants who received at least 1 full dose of VRC01 or Placebo and underwent ATI.
Measure: Median (Full Range); unit: copies/mL
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 13 | 5
copies/mL
  HIV-1 RNA at first detection | 105 [21 to 900] | 1015 [229 to 7395]
  HIV-1 RNA at ART resumption | 3440 [1587 to 31807] | 3845 [1401 to 26865]
Statistical Analysis 1: Comparison: VRC01 vs Placebo for VRC01; Test type: Superiority; p = 0.027, Wilcoxon (Mann-Whitney) — This is a p-value, comparing HIV-1 RNA levels at first detection between arms
Statistical Analysis 2: Comparison: VRC01 vs Placebo for VRC01; Test type: Superiority; p = 0.588, Wilcoxon (Mann-Whitney) — This is p-value, comparing HIV-1 RNA levels at ART resumption between arms

5. Secondary Outcome: Time to ART Resumption for Any Reason After Cessation of ART
Description: This is the days from ATI to ART resumptions.
Time Frame: Measured from Baseline ATI through ART resumption.
Population: Participants who received at least one full dose of VRC01 or placebo and underwent ATI.
Measure: Median (Full Range); unit: days
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 13 | 5
days | 35 [14 to 309] | 23 [16 to 35]
Statistical Analysis 1: Comparison: VRC01 vs Placebo for VRC01; Test type: Superiority; p = 0.031, Log Rank

6. Secondary Outcome: Number of Participants With Detectable HIV-1 RNA Via Single Copy Assay
Description: This is number of participants who had detectable HIV-1 RNA via the ultrasensitive single copy assay prior to detectability on the routine assay.
Time Frame: Measured from Baseline ATI through ART resumption.
Population: Participants who received at least 1 full dose of VRC01 or Placebo and underwent ATI.
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 13 | 5
Participants | 8 | 3

7. Secondary Outcome: Change in CD4+ T Cell Count From ATI to ART Resumption
Description: This is change in CD4+ T cell count from ATI to ART resumption.
Time Frame: Measured from Baseline ATI through ART resumption
Population: Participants who received at least 1 full dose of VRC01 or Placebo and underwent ATI.
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 13 | 5
cells/mm^3 | -37 [-258 to 101] | -21 [-248 to 258]
Statistical Analysis 1: Comparison: VRC01 vs Placebo for VRC01; Test type: Superiority; p = 0.693, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Total HIV DNA in the Peripheral Compartment
Description: This is total HIV DNA levels at baseline ATI, ART resumption and 6 month after ART resumption
Time Frame: Measured from ATI through 6 months after ART resumption
Population: Participants who received at least 1 full dose of VRC01 or Placebo and underwent ATI.
Measure: Median (Full Range); unit: copies/10^6 CD4 T cells
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 13 | 5
copies/10^6 CD4 T cells
  Total HIV DNA at baseline ATI | 16 [0 to 75] | 3 [0 to 54]
  Total HIV DNA at ART resumption | 24 [3 to 265] | 39 [5 to 169]
  Total HIV DNA at 6 months after ART resumption | 9 [0 to 56] | 15 [0 to 60]
Statistical Analysis 1: Comparison: VRC01; A comparison of total HIV DNA at baseline ATI and ART resumption within the VRC01 arm; Test type: Superiority; p = 0.15, Wilcoxon signed-rank test — The p-value is not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Placebo for VRC01; A comparison of total HIV DNA at baseline ATI and ART resumption within the placebo arm; Test type: Superiority; p = 0.04, Wilcoxon signed-rank test — The p-value is not adjusted for multiple comparisons
Statistical Analysis 3: Comparison: VRC01; A comparison of total HIV DNA at ART resumption and 6 months after ART resumption within the VRC01 arm; Test type: Superiority; p = 0.002, Wilcoxon signed-rank test — The p-value is adjusted for multiple comparisons
Statistical Analysis 4: Comparison: Placebo for VRC01; A comparison of total HIV DNA at ART resumption and 6 months after ART resumption within the placebo arm; Test type: Superiority; p = 0.22, Wilcoxon signed-rank test — The p-value is adjusted for multiple comparisons
Statistical Analysis 5: Comparison: VRC01; A comparison of total HIV DNA atbaseline ATI and 6 months after ART resumption within the VRC01 arm; Test type: Superiority; p = 0.05, Wilcoxon signed-rank test
Statistical Analysis 6: Comparison: Placebo for VRC01; A comparison of total HIV DNA at baeline ATI versus 6 months after ART resumption in the placebo arm; Test type: Superiority; p = 0.22, Wilcoxon signed-rank test

9. Secondary Outcome: Number of Participants Hospitalized.
Description: Participants were monitored for up to 10 weeks after the last infusion of VRC01 or placebo
Time Frame: Measured up to 10 weeks after the last infusion of VRC01 or placebo
Population: Participants who have been randomized to receive VRC01 or Placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 14 | 5
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Acute Retroviral Syndrome (ARS)
Description: This is the number of participants who have developed during ATI.
Time Frame: Measured from Baseline ATI through ART resumption.
Population: Participants who received at least one full dose of VRC01 or Placebo and underwent treatment interruption.
Measure: Count of Participants; unit: Participants
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 13 | 5
Participants | 0 | 0

11. Secondary Outcome: Neuropsychological Battery Performance
Description: This is a NPZ-4 score,a 4-test NP battery evaluated fine motor function/manual dexterity [Grooved Pegboard test (GP), non-dominant hand], psychomotor speed [Color Trails 1 (CT1), Trail Making A (TM)], and executive function/set shifting [Color Trails 2 (CT2)]. Individual test raw scores were converted to z-scores. Z-scores range from -3 standard deviations up to +3 standard deviations. Higher scores indicate better test performance and lower cognitive impairment.
Time Frame: Measured from Baseline ATI through ART resumption.
Population: Participants who received at least one full dose of VRC01 or Placebo and underwent ATI.
Measure: Median (Full Range); unit: Z-score
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 13 | 5
Z-score
  NPZ-4 at baseline ATI | 0.87 [0.26 to 1.48] | 1.19 [0.16 to 1.30]
  NPZ- at ART resumption | 1.25 [0.02 to 1.70] | 1.04 [0.41 to 1.73]
Statistical Analysis 1: Comparison: VRC01 vs Placebo for VRC01; Comparison between arms at baseline ATI; Test type: Superiority; p = 0.961, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: VRC01 vs Placebo for VRC01; Comparison between arms at ART resumption; Test type: Superiority; p = 0.805, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: VRC01; Comparison between Baseline and ART resumption within VRC01 arm; Test type: Superiority; p = 0.221, Wilcoxon signed-rank test
Statistical Analysis 4: Comparison: Placebo for VRC01; Comparison between Baseline and ART resumption within Placebo arm; Test type: Superiority; p = 0.500, Wilcoxon signed-rank test

12. Secondary Outcome: Computed Score on the Control and Attention Task (i.e., Flanker Task)
Description: The Flanker is a measure of executive function, specifically tapping inhibitory control and attention.The scores range from 0 to 10. A higher scores indicate higher levels of ability to attend to relevant stimuli and inhibit attention from irrelevant stimuli.
Time Frame: Measured from Baseline ATI through ART resumption.
Population: Participants who received at least 1 full dose of VRC01 or Placebo and underwent ATI.
Measure: Median (Full Range); unit: score
Arm/Group | VRC01 | Placebo for VRC01
Number analyzed (Participants) | 13 | 5
score
  Baseline ATI | 8.24 [7.43 to 9.23] | 8.36 [8.05 to 8.83]
  ART resumption | 8.4 [7.3 to 9.7] | 8.41 [7.46 to 9.18]
Statistical Analysis 1: Comparison: VRC01 vs Placebo for VRC01; Comparison between groups at baseline ATI; Test type: Superiority; p = 0.522, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: VRC01 vs Placebo for VRC01; A comparison between groups at ART resumption; Test type: Superiority; p = 0.961, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: VRC01; A comparison between baseline ATI and ART resumption within VRC01 group; Test type: Superiority; p = 0.002, Wilcoxon signed-rank test
Statistical Analysis 4: Comparison: Placebo for VRC01; A comparison between baseline ATI and ART resumption within Placebo group; Test type: Superiority; p = 0.043, Wilcoxon signed-rank test

ADVERSE EVENTS:
Time Frame: Infusion-related and unrelated Adverse Events were collected during the first study agent administration through 175 days after the last study agent administration.
Arm/Group | VRC01 | Placebo for VRC01
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/5
Other Adverse Events (participants affected / at risk) | 14/14 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VRC01 (N=14) | Placebo for VRC01 (N=5)
Fatigue (General disorders) | 7 (8) | 3 (4)
Nausea (Gastrointestinal disorders) | 5 (7) | 1 (1)
Infusion site pain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Headche (Nervous system disorders) | 4 (9) | 4 (8)
Infusion site bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Infusion site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Generalized urticaria (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1)
ALT increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal gas (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Allergy (Immune system disorders) | 1 (1) | 0 (0)
Aphthous mouth ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Chlamydia (Infections and infestations) | 0 (0) | 1 (1)
Common cold (Infections and infestations) | 1 (1) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dermatitis of dorsum, both hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Loose stool (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lymphadenopathy, right cervical (Immune system disorders) | 1 (1) | 0 (0)
Mouth sore (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Pharyngitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Syphilis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Sore throat (Gastrointestinal disorders) | 1 (1) | 1 (1)
Subconjunctival hematoma (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT02664415/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT02664415/SAP_001.pdf